CLINICAL TRIAL: NCT03623022
Title: Effects of 20,000 EU of Clinical Center Reference Endotoxin (CCRE) Versus Placebo on Systemic and Cardiovascular Inflammatory Responses in Mild Asthmatics and Healthy Volunteers
Brief Title: Effects of 20,000 EU of Clinical Center Reference Endotoxin (CCRE) Versus Placebo(ENDOHEART)
Acronym: Endoheart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); RTI International (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 17-3351
Record Dates: First submitted 2018-08-06; First posted 2018-08-09 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: healthy
MeSH Terms: interventions — Endotoxins; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects will undergo an exposure to inhaled endotoxin in a crossover fashion with normal saline inhalation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy will in charge of the randomization key, all others are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Endotoxin, then Normal Saline (Experimental): Endotoxin challenge: Subjects will undergo inhalation of 20,000 EU CCRE. The Clinical Center Reference Endotoxin (CCRE) will be inhaled by subjects as a nebulized preparation using an ultrasonic nebulizer until the challenge solution is completely spent (generally 10 minutes).
  Following a washout of 2 weeks to 3 months the participant will undergo a Saline Challenge: Subjects will undergo inhalation of 0.9% sodium chloride. The Normal saline will be inhaled by subjects as a nebulized preparation using an ultrasonic nebulizer until the challenge solution is completely spent (generally 10 minutes).
  Interventions: Drug: Clinical Center Reference Endotoxin (CCRE); Drug: Normal saline
- Normal Saline, then Endotoxin (Experimental): Saline Challenge: Subjects will undergo inhalation of 0.9% sodium chloride. The Normal saline will be inhaled by subjects as a nebulized preparation using an ultrasonic nebulizer until the challenge solution is completely spent (generally 10 minutes).
  Following a washout of 2 weeks to 3 months the participant will undergo an Endotoxin challenge: Subjects will undergo inhalation of 20,000 EU CCRE. The CCRE will be inhaled by subjects as a nebulized preparation using an ultrasonic nebulizer until the challenge solution is completely spent (generally 10 minutes).
  Interventions: Drug: Clinical Center Reference Endotoxin (CCRE); Drug: Normal saline

INTERVENTIONS:
Drug: Clinical Center Reference Endotoxin (CCRE) — subjects will undergo an exposure to inhaled endotoxin through a nebulizer for approximately 10 minutes.
  Other Names: Endotoxin
Drug: Normal saline — subjects will undergo an exposure to inhaled normal saline through a nebulizer for approximately 10 minutes
  Other Names: 0.9% sodium Chloride (NACL)

SUMMARY:
To determine the systemic inflammatory effects of inhaled endotoxin and associated alterations in cardiovascular function. Subjects will undergo an exposure to inhaled endotoxin in a crossover fashion with normal saline inhalation. Blood samples and sputum samples will be taken before and after inhalation challenge to measure markers of systemic inflammation. Cardiovascular measures, including a heart rate variability monitor, flow mediated dilation of the brachial artery and left ventricular stain will also be measured.

DETAILED DESCRIPTION:
The purpose of this study is to determine the systemic inflammatory effects of inhaled endotoxin and associated alterations in cardiovascular function. The investigators have previously found that inhalation of 20,000 Endotoxin Units (EU) of CCRE increases the neutrophil content of the blood; this dose can then be employed to screen populations for enhanced susceptibility to the systemic and cardiovascular inflammatory effect of inhaled endotoxin. Endotoxin is a commonly encountered bioaerosol and component of particulate matter (PM), a prevalent indoor and outdoor air pollutant [1-3]. For reasons that remain unclear, some individuals appear to be more susceptible to the inflammatory effects of inhaled endotoxin than are others, possibly owing to single nucleotide polymorphisms in the Toll-like receptor 4 (TLR4) gene that influence TLR4 signaling and function [4-6]. Exposure to PM is associated with increased cardiovascular morbidity and mortality [7]. PM exposure has been specifically linked with increases in blood pressure [8,9]. Susceptible individuals represent a population of particular interest for further mechanistic studies of the effects of endotoxin and for therapeutic trials. Systemic inflammatory response to inhaled endotoxin will be determined by measuring change in peripheral blood neutrophil counts, a biomarker of systemic inflammation, following inhaled CCRE vs placebo. Blood pressure, heart rate variability (HRV), vascular stiffness (by flow mediated dilation, or FMD) and left ventricular strain (LVS) will be measured before and after CCRE or placebo exposure to investigate the effect of endotoxin-induced systemic inflammation on cardiovascular function.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers with no more than mild asthma
* Age 18-50 years, inclusive, of both sexes
* Demonstrate an increase in peripheral blood PMNs of 20% (compared to baseline values) following inhalation of 20,000 EU of CCRE.
* Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy
* Normal lung function, defined as (NHanes III predicted set):

  1. Forced Vital Capacity (FVC) of > 80 % of that predicted for gender, ethnicity, age and height
  2. Forced Expiratory Volume in the first second of the exhale (FEV1) of > 80 % of that predicted for gender, ethnicity, age and height
  3. FEV1/FVC ratio of > .75 of that predicted for gender, ethnicity, age and height
* Oxygen saturation of > 93%, and blood pressure within the following limits: (Systolic between 150 - 90, Diastolic between 90-60 mm Hg)

Exclusion Criteria:

* Any chronic medical condition considered by the PI as a contraindication to the exposure study including significant cardiovascular disease, diabetes requiring medication, chronic renal disease, or chronic thyroid disease.
* Physician directed emergency treatment for asthma exacerbation within the preceding 3 months.
* Exacerbation of asthma more than 2x/week that would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma.
* Nighttime symptoms of cough or wheeze greater than 1x/week at baseline (not during a clearly recognized viral induced asthma exacerbation) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma
* Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness) which would be characteristic of a person of moderate or severe persistent asthma as outlined in the current NHLBI guidelines for diagnosis and management of asthma. (Not to include prophylactic use of albuterol prior to exercise).
* History of intubation for asthma
* Daily use of NSAIDs, or inability to withhold NSAIDs for 4 days prior to dosing.
* Use of medications that may impact the results of the study to include, but not limited to, systemic corticosteroids, beta blockers.
* Cigarette smoking > 1 pack per month.
* Body Mass Index >35 kg/m2.
* Pregnant or breast feeding women
* Subjects who are employed within the past 6 months in an occupation with high risk for endotoxin exposure, such as grain storage sites or swine containment.
* Any acute, non-chronic medical condition requiring treatment, such as bronchitis, pneumonia or febrile illness within the prior 4 weeks.
* Participation in studies involving new molecular entities or an experimental environmental exposure in the past 4 weeks.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular Strain | 15 minutes and 4 hrs after inhalation
  Comparing pre and post results before and after endotoxin vs normal saline inhalations
Change in Flow Mediated Dilation | 15 minutes and 4 hrs after inhalation
  Comparing pre and post results before and after endotoxin vs normal saline inhalations

SECONDARY OUTCOMES:
Percent Change in sputum Polymorphonuclear Neutrophils (PMNs) | 6 hrs after inhalation
  post differences in % change comparing saline to endotoxin
Percent Change in Blood Polymorphonuclear Neutrophils (PMNs) | 5 hours and 30 minutes after inhalation
  post differences in % change comparing saline to endotoxin

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No